CLINICAL TRIAL: NCT01614236
Title: Pre- Versus Post-Incisional Pregabalin for Postoperative Pain Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Michal Roll PhD,MBA, Resarch and developement Director, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TASMC-08-WAA-024811-TLV
Record Dates: First submitted 2012-06-03; First posted 2012-06-07 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Postoperative Pain Control; Multimodal Analgesia
Keywords: pregabalin; analgesia; postoperative pain; orthopedic oncology patients
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Pregabalin; Injections, Epidural

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Active Comparator): patients will be randomized similarly but will undergo surgery under epidural analgesia
  Interventions: Drug: epidural
- Lyrica (Active Comparator): Patients will received 150 mg of PGL or placebo at 20:00 the evening before surgery and 1.5 h before surgery and will undergo surgery under GA
  Interventions: Drug: pregabalin

INTERVENTIONS:
Drug: pregabalin — Patients in one set (40 patients/sct) will received 150 mg of PGL or placebo at 20:00 the evening before surgery and 1.5 h before surgery and will undergo surgery under GA
  Arms: Lyrica
Drug: epidural — patients will be randomized similarly but will undergo surgery under epidural analgesia
  Arms: control

SUMMARY:
Proper pain relief is a major concern of patients worldwide. Preoperatively, one of the most common questions asked by patients pertains to the amount of pain they will experience after surgery how long it will last and how good will it be controlled. Pain concerns the surgical team as well, because of its correlation with clinical outcomes and patients' satisfaction rate . Studies have shown that negative clinical outcome with regard to pain control includes decreases in vital capacity and alveolar ventilation, pneumonia, tachycardia, hypertension, myocardial ischemia, transition into chronic pain, poor wound healing, and psychological sequelae .

DETAILED DESCRIPTION:
Pregablain Interest has been focused on the analgesic, sedative, anxiolytic, and opioid¬sparing effects of pregabalin (PGL) (S+ 3-isobutyl GABA), a structural analog of GABA and a derivative of gabapentin in various pain settingsl including postoperative pain . Of a similar mechanism of action, it is thought to possess a superior phannacokinetic profile than gabapentin [15]. Pregabalin has a variable role in neuropathic pain conditions, such as post-herpetic neuralgia, painful diabetic neuropathy, central neuropathic pain, and fibromyalgia . Some studies had not demonstrated a significant analgesic effect in the acute, postoperative pain; others propose PGL to have effective sedative and opioid-sparing effects, both useful characteristics for the control of acute pain. Opioid sparing effects and improved pain scores have been seen after abdominal and pelvic surgery. Its many potential actions such as reducing opioid reqUirements, prevention and reduction of opioid tolerance, improvement of the quality of opioid analgesia, decreased respiratory depression, relief of anxiety, and gastriC sparing, make it an attractive drug to consider for control of pain in the post operative period.

Population characteristics The orthopedic oncological patients are a specific group of individuals whose demand for antinociception starts rather before surgery because of the bone tumor-generated pain that usually signals the first the existence of pathology. Also, pain intensity that is generated by an intervention on the skeleton is more intense than that induced by damage to soft tissue. Subsequently, these patients would require postoperatively more analgesics than after general surgery and for a longer period of time. We have demonstrated previously that acute pain that is superimposed on an already aroused eNS, i.e., the presence of central sensitization, would create a situation where complete antinociception is hard to obtain, as in these patients, and therefore the efficacy of the antinociceptive protocol is best tested, comprised the possible transformation of acute into chronic pain.

Pre-emption has been pointed out as a beneficial tool for reducing perioperative pain. Various techniques have been employed for this purpose; different drugs were used as well. The beneficial effects of preemptive PGL were documented in patients who had undergone lumbar discectomy, both immediately and 1 and 3 months after surgery.

Hypothesis No studies considered the comparison of preemptive vs. post-surgery PGL only administration, We believe that the administration of PGL preemptively would diminish pain sensation and therefore the need for opioids administration in orthopedic-oncologic patients more effectively than if administered starting postoperatively.

Objectives To assess the beneficial effects Of PGL admi"istered either pre-incisionally or post-incisionally on the immediate and late (1-and 3 months) postoperative analgeSia requirements and pain scores, as well as satisfaction rate in the orthopedic oncologic patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA phYSical status I-III patients who will undergo bone with or without soft tissue cancer surgery type II and III under general or epidural anesthesia

Exclusion Criteria:

* Allergy to opioids, bupivacaine, midazolam, PGL, or non¬steroidal anti-infiammatory dnugs (NSAIDs)
* History of chronic pain or psychiatric disorders
* Use of centrally acting drugs of any sort.
* Soldiers and pregnant women will also be excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
post-operative pain score | 4 days

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel